CLINICAL TRIAL: NCT06556485
Title: Preventive Catheter Ablation for Ventricular arrhythmiaS in Patients With End-sTage Heart faiLure rEfferred for Heart Transplantation eValuaTion (CASTLE-VT)
Brief Title: Preventive Catheter Ablation for Ventricular arrhythmiaS in Patients With End-sTage Heart faiLure
Acronym: CASTLE-VT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDZ-ER_004_CS
Record Dates: First submitted 2024-07-17; First posted 2024-08-16 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure; Arrhythmia, Ventricular; Cardiomyopathy Ischemic; Catheter Ablation; Heart Transplantation; Left Ventricular Assist Device
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac | interventions — Catheter Ablation; Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ablation group (Active Comparator): Primary prophylactic ablation
  Interventions: Procedure: Catheter ablation
- Control group (Active Comparator): Optimal medical therapy
  Interventions: Drug: Medical therapy

INTERVENTIONS:
Procedure: Catheter ablation — Preventive ablation therapy
  Other Names: Ablation
  Arms: Ablation group
Drug: Medical therapy — Optimal medical therapy
  Other Names: Medical
  Arms: Control group

SUMMARY:
CASTLE-VT is a randomized evaluation of prophylactic ablative treatment of arrhythmogenic ventricular scar in patients referred for HTx evaluation and diagnosed with ICM. Ablation will be performed with the use of a substrate-based approach in which the myocardial scar is mapped and ablated while the heart remains predominantly in sinus rhythm. The primary end point is the composite of all-cause mortality, worsening of HF requiring prioritized transplantation or LVAD implantation. The main secondary study end points are all-cause mortality, cardiovascular mortality, incidence of implantable cardioverter-defibrillator (ICD) therapy, hospitalizations, Quality of life, time to first ICD therapy, number of device-detected ventricular tachycardia/ventricular fibrillation episodes, LV function, and exercise tolerance. CASTLE-VT will randomize 160 patients with a follow up period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic cardiomyopathy with left ventricular ejection fraction ≤ 35% (measured in the last 6 weeks prior to enrollment)
2. Eligible for heart transplantation due to end-stage heart failure
3. NYHA class ≥ III
4. Impaired functional capacity or inability to exercise
5. Indication for ICD therapy due to primary prevention
6. Implanted ICD or ICD implantation within 3 months after randomization
7. The patient is willing and able to comply with the protocol and has provided written informed consent
8. Age ≥ 18 years

Exclusion Criteria:

1. Previous catheter ablation for ventricular arrhythmias
2. Previous appropriate ICD-therapy for ventricular arrhythmias
3. Acute coronary syndrome, cardiac surgery, angioplasty, or cerebrovascular accident within 4 weeks prior to enrollment
4. Untreated hypothyroidism or hyperthyroidism
5. Woman currently pregnant, breastfeeding, or not using reliable contraceptive measures during fertility age
6. Mental or physical inability to participate in the study
7. Listed as "high urgent" for heart transplantation
8. Cardiac assist device implanted
9. Planned cardiovascular intervention
10. Life expectancy ≤ 12 month
11. Uncontrolled hypertension
12. Requirement for dialysis due to end-stage renal failure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary end point | through study completion, an average of 2 years
  Composite of all-cause mortality, worsening of HF requiring prioritized transplantation or LVAD implantation

SECONDARY OUTCOMES:
Secondary end point 1 | through study completion, an average of 2 years
  all-cause mortality, cardiovascular mortality
Secondary end point 2 | through study completion, an average of 2 years
  incidence of implantable cardioverter-defibrillator (ICD) therapy, hospitalizations, number of device-detected ventricular tachycardia/ventricular fibrillation episodes
Secondary end point 3 | through study completion, an average of 2 years
  Quality of life, time to first ICD therapy
Secondary end point 4 | through study completion, an average of 2 years
  LV function, exercise tolerance

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Electrophysiology, Herz- und Diabeteszentrum NRW, Bad Oeynhausen, Germany